CLINICAL TRIAL: NCT04029727
Title: Pilot Study to Evaluate the Effect of the Consumption of a Combination of Plant Extracts (BSL_EP025) on the Levels of LDL-cholesterol and Oxidized LDL-cholesterol in Healthy Volunteers
Brief Title: Effect of the Combination of Plant Extracts (BSL_EP025) in Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C025
Record Dates: First submitted 2019-07-22; First posted 2019-07-23 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Disease
Keywords: Plant extract; LDL cholesterol; Dietary supplement
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of Plant Extracts (BSL_EP025) (Experimental): The volunteers will take two capsules daily with a combination of plant extracts (BSL_EP025)
  Interventions: Dietary Supplement: Combination of Plant Extracts (BSL_EP025)
- Placebo (Placebo Comparator): The volunteers will take two capsules daily with maltodextrin.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Combination of Plant Extracts (BSL_EP025) — Each participant will consume 2 capsules daily at lunch for 8 weeks.
  Arms: Combination of Plant Extracts (BSL_EP025)
Dietary Supplement: Placebo — Each participant will consume 2 capsules daily at lunch for 8 weeks.
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the ability of a combination of plant extracts (BSL_EP025) to reduce the levels of LDL-cholesterol and oxidized LDL-cholesterol in individuals with LDL-cholesterol levels between 100 and 190 mg/dL.

DETAILED DESCRIPTION:
There is a strong relationship between serum cholesterol levels and cardiovascular diseases, especially between coronary artery disease and LDL-cholesterol (LDL).

LDL is the lipoprotein responsible for delivering cholesterol to cells. However, in recent years, special attention has been given to modified LDL, especially oxidized LDL, since it plays a very important role in the initiation and progression of the atheroma plaque.

There are environmental and genetic factors that can influence the type and levels of blood lipoproteins. Among the modulable factors (environmental) it has been observed that some phytochemical compounds found in several plant extracts may reduce cardiovascular risk, due to their antioxidant and anti-inflammatory properties.

The objective of the present study is to evaluate the possible effect of the intake of a combination of plant extracts (BSL_EP025) on the levels of LDL-cholesterol and oxidized LDL-cholesterol in healthy individuals with LDL-cholesterol levels between 100 and 190 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 65 years of age.
* Levels of LDL-cholesterol between 100 and 190 mg/dL.
* Accept freely to participate in the study and sign the informed consent document.

Exclusion Criteria:

* Be pregnant.
* Have planned to carry out a dietary intervention or exercise practice with the aim of losing weight in the coming weeks.
* Suffer from a serious illness.
* Have diabetes.
* Having a cerebrovascular disease.
* Be taking products or drugs to control cholesterol levels or with antioxidant activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 8 weeks
  Levels of LDL cholesterol in plasma
Oxidized LDL cholesterol | 8 weeks
  Levels of oxidized LDL cholesterol in plasma

SECONDARY OUTCOMES:
Total cholesterol | 8 weeks
  Levels of total cholesterol in plasma
HDL cholesterol | 8 weeks
  Levels of HDL cholesterol in plasma
Triglycerides | 8 weeks
  Levels of triglycerides in plasma
Glucose | 8 weeks
  Levels of glucose in plasma
Blood pressure | 8 weeks
  Systolic and diastolic blood pressure
Body mass index | 8 weeks
  Weight/height ratio
VCAM-1 | 8 weeks
  Plasma levels of VCAM-1
ICAM-1 | 8 weeks
  Plasma levels of ICAM-1
Beta IL-1 | 8 weeks
  Plasma levels of beta IL-1
IL-6 | 8 weeks
  Plasma levels of IL-6
IL-10 | 8 weeks
  Plasma levels of IL-10

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Quesada, MD, PhD, Study Chair — Medical specialist in Endocrinology, Hospital San Cecilio de Granada
Locations (1):
- Biosearch Life, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No